CLINICAL TRIAL: NCT04405895
Title: Effect Meal Timing in Type 2 Diabetes on Serum Induced SIRT1 and Clock Gene Expression in Hepatocytes
Brief Title: Effect of Meal Timing in T2D on Hepatocytes SRIT1 and Clock Genes
Acronym: Liver-CG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Daniela Jakubowicz, MD: Clinical Profesor Head of Obesity Clinic at Diabetes Unit., Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0118-20-WOMC
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Diabetes; Meal Timing; Clock Genes; Hepatocytes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The researcher will explore the effect of serum samples collected from T2D participants following either Breakfast Diet (3Mdiet) or Allday Diet (6Mdiet) schedule, on SIRT1 and Clock Gene circadian expression of cultured hepatocytes using the ex-vivo/in-vitro approach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast Diet (3Mdiet) (Experimental): The Breakfast Diet (3Mdiet) will consist in 3 meals with distribution of calories: breakfast 50%, lunch 33% and dinner 17%.
  Interventions: Other: Breakfast Diet
- Allday Diet (6Mdiet) (Active Comparator): The Allday Diet (6Mdiet) will consist on 6 meals (breakfast, lunch and dinner and 3 snacks) with distribution of calories: breakfast 15%, lunch 25%, dinner 30% and 10% in each of the three snacks.
  Interventions: Other: Allday Diet

INTERVENTIONS:
Other: Breakfast Diet — Breakfast Diet (3Mdiet) consist on high-energy breakfast and reduced in energy and carbohydrate (CH) dinner. Participants fasting serum to provide serum to for the in ex-vivo cell studies, will be collected at fasting (8:00), at start (day 0), after 2 weeks and at the end of 3Mdiet intervention (12 weeks). The participants serum is added to culture medium (as serum conditioned medium) to treat during 48 hours the cultured hepatocytes. After 48 hours of serum treatment, the mRNA extraction for the assessment of SIRT1 and Clock Gene expression will be performed at 00:00, 06:00, 12:00 and at 18:00 to assess SIRT1 and the Clock Genes circadian oscillation in hepatocytes. The 3Mdiet efficacy on reducing the overall glycemic excursions is assessed with continuous monitoring system at baseline after 2 weeks month of diet intervention.
  Other Names: 3Mdiet
  Arms: Breakfast Diet (3Mdiet)
Other: Allday Diet — Allday Diet (6Mdiet) consist in 6 small meals: breakfast, lunch and dinner and 3 snacks, with calories and carbohydrates (CH) evenly distributed throughout the day. Participants fasting serum to provide serum to for the in ex-vivo cell studies, will be collected at fasting (8:00), at start (day 0), after 2 weeks and at the end of 6Mdiet intervention (12 weeks). The participants serum is added to culture medium (as serum conditioned medium) to treat during 48 hours the cultured hepatocytes. After 48 hours of serum treatment, the mRNA extraction for the assessment of SIRT1 and Clock Gene expression will be performed at 00:00, 06:00, 12:00 and at 18:00 to assess SIRT1 and the Clock Genes circadian oscillation in hepatocytes. The 6Mdiet efficacy on reducing the overall glycemic excursions is assessed with continuous monitoring system at baseline after 2 weeks month of diet intervention.
  Other Names: 6Mdiet
  Arms: Allday Diet (6Mdiet)

SUMMARY:
This study is undertaken to explore in T2D, the effect of meal timing on serum induced SIRT1 and Clock Genes mRNA expression in cultured hepatocytes. Fasting serum samples were collected from T2D participants, following two different meal timing schedules, either a diet with large breakfast and lunch with small dinner Breakfast Diet (3Mdiet) or an isocaloric diet with 6 small meals evenly distributed along the day Allday Diet (6Mdiet). The researchers will use an ex-vivo/in-vitro approach in which cultured medium will be conditioned with the fasted human serum collected from the two groups of T2D participants at baseline, after 2 weeks and after 12 week of the diet intervention.

DETAILED DESCRIPTION:
The timing of many physiological processes, including glucose metabolism, is coordinated by the circadian clock gene system. The circadian clock regulation, optimize glucose metabolism for the consumption of high energy and carbohydrate (CH) meals in the early hours of the day and for fasting at evening and night. Circadian disruption which occurs when the meal timing is not aligned with the circadian clock rhythms like skipping breakfast, overeating CH at night or eating CH all day, lead to desynchronized clock genes and can result in adverse health outcomes like insulin resistance, obesity hyperglycemia and T2D. Although the clock genes are disseminated in almost all peripheral tissues, those localized in the liver, are particularly important for the regulation of glucose metabolism, influencing the enzymatic determinants of the hepatic glucose output, by enhancing glycogen storage and suppressing nocturnal hepatic glucose production (glycogenolysis and gluconeogenesis sequentially).Therefore, the disruption of the hepatic clock genes lead to fasting, nocturnal, and to postprandial hyperglycemia in T2D. The researchers had previously shown in T2D, that compared to 6Mdiet, the 3Meal diet timing schedule, was most effective in reducing body weight, HbA1c, overall hyperglycemia, and led to up-regulation of SIRT1 and Clock Genes mRNA expression in leukocytes. However, this effect of meal timing had never been explored in liver cells. The investigators hypothesized that compared to Allday Diet (6Mdiet), the serum collected from T2D participants following Breakfast Diet (3Mdiet) will up-regulate SIRT1 and Clock Genes oscillatory mRNA expression in cultured hepatocytes.

ELIGIBILITY:
Inclusion Criteria:

* T2D patients with stable treatment for at least 3 month preceding the study.
* HgA1c >7.5 %.
* Age > 30 years.
* BMI: 27-34 kg/m2.
* Treatment with antidiabetic drugs (i.e. metformin, DPP4 inhibitors, glinides) and GLP-1 analogs, will be allowed
* Anti-hypertensive treatment will be allowed.
* Lipid-lowering medication also allowed

Exclusion Criteria:

* Type 1 diabetes.
* Major illnesses (liver, heart, kidney, infectious, neurological, psychiatric, immunological, active malignancy).
* Change in weight of > 4.5 kg within 3 month prior the diet onset.
* Night or rotating shift workers.
* Those who crossed more than 2 time zones during 2-week period prior to study onset.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-05-31 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in Clock Genes mRNA | Baseline and at 2 weeks post diet intervention
  Change from baseline serum-induced hepatocyte Clock Gene mRNA expression, will be assessed at 2 weeks post diet intervention in the two groups:Breakfast Diet (3Mdiet) and Allday Diet (6Mdiet)

SECONDARY OUTCOMES:
Change in Clock Genes expression | Baseline and at 12 weeks post diet intervention
  Change from baseline serum-induced hepatocyte Clock Gene expression, will be assessed at 12 weeks post diet intervention in the two groups: Breakfast Diet (3Mdiet) and Allday Diet (6Mdiet)
Change in SIRT1 mRNA expression | Baseline and at 2 weeks post diet intervention
  Change from baseline serum-induced hepatocyte SIRT1 mRNA expression, will be assessed at 2 weeks post diet intervention in the two groups: Breakfast Diet (3Mdiet) and Allday Diet (6Mdiet)
Change in Overall Glycemia | Baseline and at 12 weeks post diet intervention
  Change from baseline in overall glycemia will be assessed at 12 weeks post diet intervention in the two groups: Breakfast Diet (3Mdiet) and Allday Diet (6Mdiet) Overall glycemia will be test by using continuous blood monitoring system

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Wolfson Medical Center; Shani Tsameret, RD, Principal Investigator — E. Wolfson Medical Center.
Locations (1):
- Wolfson Medical Center, Holon, Please Select, Israel